CLINICAL TRIAL: NCT00678054
Title: A Phase II Study of Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF) for the Treatment of Patients With Evidence of Serologic (PSA) Progression After Definitive Therapy for Localized Prostate Cancer
Brief Title: Study of Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF) for Patients With Rising Prostate-Specific Antigen (PSA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCSF99551
Record Dates: First submitted 2008-02-20; First posted 2008-05-15 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF) (Experimental)
  Interventions: Drug: GM-CSF

INTERVENTIONS:
Drug: GM-CSF — Each cycle will consist of 28 days. Patients will receive 250 ug/m2/day of GM-CSF administered subcutaneously on days 1-14.

SUMMARY:
This is a Phase II study to test the efficacy of exogenously administered GM-CSF in prostate cancer patients who have failed definitive local therapy, and have only serologic (PSA) evidence of progression.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of adenocarcinoma of the prostate; stage T1-T3, N0-N1, M0
* Prior definitive therapy for primary prostate cancer consisting of:external beam radiotherapy;brachytherapy with or without pelvic external beam radiation; or radical prostatectomy with or without adjuvant or salvage radiation therapy
* Therapeutic PSA response to primary therapy below 1.0 ng/ml post radiation therapy or below 0.4 ng/ml for radical prostatectomy
* Patients treated with adjuvant or salvage radiation therapy following radical prostatectomy are eligible provided:Post prostatectomy PSA was never > 6.0 ng/ml, last effective day of androgen deprivation is at least 3 months prior to study entry
* Recurrent PSA level elevation (between 0.4 ng/ml and 6.0 ng/ml) on two determinations at least one week apart.
* No clinical evidence of gross local recurrence or known metastatic disease other than PSA elevation. Transrectal ultrasound and/or biopsy to evaluate local recurrence is not required. All patients will receive a bone scan and CT scan of the abdomen to exclude metastases.
* Estimated life expectancy of at least 6 months.
* ECOG Performance status of 0 or 1.
* Willing and able to give informed consent.

Exclusion Criteria:

* Cryosurgery as definitive therapy of primary tumor.
* Any metastasis.
* No concurrent or prior malignancy is allowed except for the following: adequately treated basal or squamous cell skin cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years.
* Current systemic steroid therapy (inhaled or topical steroids acceptable).
* Prior hormonal therapy for treatment of progressive disease.
* Prior chemotherapy, immunotherapy, or therapy with other experimental agents for prostate cancer.
* Any surgery within the prior 4 weeks.
* Bilirubin and SGOT > 2 x upper limit of normal.
* BUN and serum creatinine > 2.0 times normal.
* No active congestive heart failure.
* If there is a history of clinically significant obstructive airway disease, a DLCO must exceed 50%.
* Active uncontrolled bacterial, viral or fungal infection until these conditions are corrected or controlled.
* Any underlying medical condition which in the principal investigator's opinion will make the administration of GM-CSF hazardous or obscure the interpretation of adverse events.
* PSA > 6.0 ng/ml

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 1999-04; Primary Completion 2000-08-11 (Actual); Study Completion 2015-10-23 (Actual)

PRIMARY OUTCOMES:
PSA Response | Monthly

CONTACTS AND LOCATIONS:
Overall Officials: Eric Small, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States

REFERENCES:
- [Result] Rini BI, Weinberg V, Bok R, Small EJ. Prostate-specific antigen kinetics as a measure of the biologic effect of granulocyte-macrophage colony-stimulating factor in patients with serologic progression of prostate cancer. J Clin Oncol. 2003 Jan 1;21(1):99-105. doi: 10.1200/JCO.2003.04.163. PMID 12506177